CLINICAL TRIAL: NCT03340896
Title: Phase III Trial of Laryngeal Preservation Comparing Induction Chemotherapy With Cisplatin, 5-fluorouracil and Docetaxel (TPF) Followed by Radiotherapy and Concomitant Administration of Radiotherapy With Cisplatin
Brief Title: Trial of Laryngeal Preservation Comparing Induced CT Followed by RT vs CT Concomitant to RT
Acronym: SALTORL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC 2014-03
Record Dates: First submitted 2016-03-08; First posted 2017-11-14 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Larynx, hypopharynx
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Laryngeal Diseases | interventions — Docetaxel; Cisplatin; Fluorouracil; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TPF followed by radiotherapy (Active Comparator): Induction chemotherapy by Docetaxel 75 mg/m² day 1,cisplatin 75 mg/m² day 1 and 5 fluorouracil 750mg/m²(day 1 to day 5) 3 cycles day1, day 22, day 43 followed (for responders or stable disease patients) by radiotherapy
  Radiotherapy ;70 gray fractionization: 2Gy/day, 5days/week, for 7 weeks.
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Drug: Fluorouracil; Radiation: radiotherapy
- Cisplatin and radiotherapy (Experimental): Drug and radiation • Cisplatin: 100 mg / m² administered IV at J1, J22 and J43 of radiotherapy
  . Radiotherapy 70 gray fractionization: 2Gy/day, 5days/week, for 7 weeks.
  Interventions: Drug: Cisplatin; Radiation: radiotherapy

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 75 mg / m² administered on day 1 of each cycle every 3 weeks as an intravenous (IV) infusion of one hour followed by cisplatin 75 mg / m² administered on day 1 hour infusion followed by 5-FU, 750 mg / m² / day administered in continuous infusion from D1 to D5 (or 120 hours)
  Other Names: Taxotere
  Arms: TPF followed by radiotherapy
Drug: Cisplatin — Cisplatin: 75 mg/m² for experimental arm and 100mg/m² for comparator arm administered on day 1 of each cycle every 3 weeks as an intravenous (IV) infusion.
  Other Names: Cisplatine
Drug: Fluorouracil — 5-FU, 750 mg / m² / day administered in continuous infusion from D1 to D5 (or 120 hours)
  Other Names: 5 FU
  Arms: TPF followed by radiotherapy
Radiation: radiotherapy — Radiotherapy : 70Gy (2Gy/day) for 7 weeks.
  Other Names: radiation therapy

SUMMARY:
This study compare the survival without laryngeal dysfunction 2 years after the end of treatment, obtained by chemotherapy followed by radiotherapy or chemotherapy with cisplatin administrated during radiotherapy.

DETAILED DESCRIPTION:
In patients with tumors classified as T3 or T4 larynx and hypopharynx, the usually recommended treatment was total laryngectomy.This intervention allows to obtain locoregional disease control in 75% of cases, without laryngectomy

TPF arm followed by radiotherapy was validated in a Phase III (GORTEC 2000-01), it will be the standard treatment.

The RTOG study concluded that chemotherapy administrated during radiotherapy became a standard of laryngeal preservation.

Taking together all these considerations, it is necessary to perform a direct comparison in a randomized trial to further test this hypothesis. Chemotherapy followed by radiotherapy will be the standard arm. It hopes to increase the survival rate from 52% to 65% in the experimental arm.

ELIGIBILITY:
Inclusion Criteria:

* Squamous cell carcinoma of the larynx or hypopharynx, histologically proven, locally advanced:

  * T2 not accessible to a supra-cricoid partial laryngectomy or not,
  * T3 without massive infiltration by endolarynx transglottic injury,
  * N0 to N2c
  * No distant metastasis
  * No associated cancer or earlier
* Patients Previously Untreated
* Age> 18 years and <75 years
* PS 0 or 1 according to WHO
* Tumor volume assessable by RECIST.
* Absence of distant metastasis, confirmed by chest TDM, abdominal ultrasound (or TDM) in case of abnormal liver function and bone scan if local symptoms.
* Absence of any participation in a clinical trial within 30 days prior to inclusion.
* Absence of any concomitant cancer treatment.
* Absence of any chronic treatment ( ≥3 months) with a daily corticosteroid dose is ≥20 mg / day of methylprednisolone or equivalent.
* Hematological function: neutrophils ≥1.5 x 109 / L, platelets ≥100 x 109 / l, hemoglobin ≥10 g / dl (or 6.2 mmol / l).
* Hepatic function: normal total bilirubin; AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN (LNS) of each center; alkaline phosphatase ≤ 5 x LNS.
* Renal function: serum creatinine ≤ 120 mol / l (1.4 mg / dl); if creatinine > 120 mol / l, creatinine clearance should be ≥ 60 ml / min.
* calculated creatinine clearance (Crockcroft formula) or measured ≥ 60 ml / min
* Estimated life expectancy ≥ 3 months
* Weight loss less than 10% over the last 3 months
* Patient has given its written consent before any specific procedure of the Protocol.
* Women and men of childbearing age should have accepted a medically effective contraception during the treatment period and at least 6 months after discontinuation of study treatments (Docetaxel, 5-Fluorouracil and Cisplatin. If pregnancy is declared by a patient or partner of a patient, it must be followed to know the evolution of pregnancy.

Exclusion Criteria:

* transglottic T3 with massive infiltration of hemilarynx or T4 with massive cartilaginous tumor lysis or reverse cricoarythénoïdenne region or posterior hypopharyngeal wall
* tumor requiring the completion of an immediately tracheotomy.
* Tumour available immediately to partial surgery.
* tumor requiring circular hypopharyngectomie
* N3 nodal injury
* Vaccination against yellow fever recent or anticipated
* Deficit known dihydropyrimidine dehydrogenase (DPD)
* Other malignancies within 5 years prior to randomization, with the exception of adequately treated basal skin cancer and carcinoma in situ of the cervix.
* Patients with AST or ALT> 1.5xULN associated with alkaline phosphatase > 2.5x LNS will not be eligible for testing.
* symptomatic neuropathy grade ≥2 with NCI-CTC.
* Clinical alteration of hearing function.
* Other concomitant serious medical conditions (partial list):

  * Unstable cardiac disease despite treatment.
  * Myocardial infarction within 6 months prior to trial entry.
  * Neurological or psychiatric history such as dementia, seizures;
  * Severe uncontrolled infection.
  * Significant gastrointestinal abnormalities, including those that require parenteral nutrition, active peptic ulcer disease and a history of surgical procedures affecting absorption
  * Obstructive pulmonary disease requiring hospitalization in the year before inclusion.
  * Unstable diabetes or other cons-indications to corticosteroids.
  * Significant ophthalmologic abnormality.
  * Moderate or severe eczema.
* Allergy to iodine.
* Hypersensitivity to Docetaxel, Cisplatin or at one of their excipients.
* Concomitant use of phenytoin, carbamazepine, barbiturates and rifampicin.
* Presence, selection, psychological factors, family, social or geographical may alter patient compliance with the study protocol and follow-up, a criterion of non-inclusion. These factors should be discussed with the patient before inclusion in the trial.
* Pregnant or nursing women.
* Patient (male or female) of childbearing age not taking adequate contraceptive measures.
* Patient deprived of their liberty, without guardianship or curatorship.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2015-06-25 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
free survival | 24 months after treatment initiation
  Minimum time between randomization and the occurrence of events such as: death, total laryngectomy, tracheotomy.

SECONDARY OUTCOMES:
Overall survival | 60 months
  "From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months").
Progression free survival | 60 months
  "From date of randomization until the date of first documented progression assessed up to 60 months").
Larynx Preservation | 24 months after treatment initiation
  From date of randomization up to 24 months evaluated by dynamic deglutition videoscopy
Feasibility of salvage surgery | 60 months after randomization
  Assessing the number of recurrences that could be successfully treated with salvage surgery and description of postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Yoann POINTREAU, Dr, Principal Investigator — Centre Jean Bernard
Locations (1):
- Centre Jean Bernard, Le Mans, France

IPD SHARING:
Plan to Share IPD: No